CLINICAL TRIAL: NCT02996929
Title: Prospective, Investigational Study to Assess the Safety and Performance of LeadExx LC System in Lead Extraction
Brief Title: Safety and Performance of LeadExx LC System in Lead Extraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LeadExx Cardiac Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Leadexx CL-001
Record Dates: First submitted 2016-12-11; First posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Implant Site Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study group (Experimental): Subjects who are scheduled for CIED lead extraction with the LC system
  Interventions: Device: LC System

INTERVENTIONS:
Device: LC System — Subjects will undergo CIED lead extraction with the LC system

SUMMARY:
The study's main purpose is to evaluate the safety and performance of the LeadExx LC System and its ability to safely extract leads.

The study will enroll 10 patients scheduled for CIED lead extraction. The decision upon lead extraction will be based upon the applicable Heart Rhythm Society guidelines or European Heart Rhythm Association (EHRA).

DETAILED DESCRIPTION:
The use of implantable cardiac devices has been exponentially increasing, and lead extraction has become a necessary procedure. But lead extraction has potentially serious complications, including venous or myocardial tear, cardiac tamponade, and even death. Powered sheaths, such as Excimer laser or a radiofrequency system, have been used for extraction of ICD or pacemaker leads. However, the Heart Rhythm Society (HRS) has stated that "possible predictors of major complications were implant duration of the oldest lead, female gender, ICD lead removal, and use of the laser extraction technique, multiple leads, and calcified leads".

To reduce the risk of the lead extraction procedure and therefore reduce the number of abandoned leads, LeadExx had developed its system.

The LC system is an active disposable system provided sterile for single use. The system is comprised of the following two main parts:

a. Dilation Unit (DU) - (invasive, sterile) b. Control Unit- (CU) - (non-invasive, sterile fluid path) The physical connection between the units is achieved by 3 Luer locks that connect the CU Solenoids' output to 3 flexible tubes at the proximal end of the DU.

1. Dilation Unit (DU):

   The dilation unit is an invasive sterile unit, comprised of a dilation tip and a connecting shaft. The unit is activated using a hydraulic mechanism.

   The dilation tip is threaded over the lead, inserted into the vessel together with its connecting shaft and while advancing along the lead, dilates the surrounding tissue and ultimately enables the lead removal from the vein.
2. Control Unit (CU):

The Control Unit is a non-invasive fluid path sterile unit, comprised of various off the shelf modules . The unit is being filled with sterile Saline just prior to its operation and by synchronizing the transfer of the Saline into the DU controls its advancement. I

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18-75 years old.
2. Scheduled for an CIED lead extraction upon current guidelines
3. Willing and able to sign the informed consent.
4. Lead implant duration more than 1 year and less than 5 years.
5. Patient with Lead size 7F
6. BMI 22-32
7. Number of implanted leads 1-3

Exclusion Criteria:

1. Lead implant duration is less than 1 year or more than 5 years.
2. Patients with acute and chronic lead infections
3. Pericardial or subcutaneous CIED systems (without trans venous CIED lead)
4. Pregnant or lactating.
5. Patients with expected survival of less than 1 year.
6. Subjects who are participating in another clinical study.
7. Subjects who are unable or unwilling to follow the study schedule of visits.
8. Contraindication to administration of iodinated contrast (creatinine > 2.0 or contrast allergy)
9. Patients with a history of venous thromboembolism, coagulopathy or malignancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 1 month
  Monitoring Adverse events that are related to the extraction procedure, or the extraction system

SECONDARY OUTCOMES:
Performance | During procedure
  Secondary Objectives:
  To assess the ease of use by questions
  * Duration of procedure,
  * Physician satisfaction by questions
Practical removal of intact lead | During procedure
  Performance primary objective:
  To verify that the attachment and advancement of the LC system enables a safe and practical removal of the Lead.

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Nof, Dr., Principal Investigator — Sheba Medical Center

IPD SHARING:
Plan to Share IPD: No